CLINICAL TRIAL: NCT00984893
Title: A Real-world Study Cohort of Postmenopausal Women With Osteoporosis Taking Zoledronic Acid or Oral Bisphosphonates
Brief Title: Intra-venous Zoledronic Acid Once Yearly
Acronym: IVORY
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CZOL446HCA10
Record Dates: First submitted 2009-09-23; First posted 2009-09-25 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Post-Menopausal Osteoporosis
Keywords: Osteoporosis; Bone Mineral density; fragility fractures; zoledronic acid.; Treatment
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Zoledronic Acid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Zoledronic acid
  Interventions: Drug: zoledronic acid
- Oral Bisphosphonates
  Interventions: Drug: Any oral bisphosphonates marketed in Canada

INTERVENTIONS:
Drug: zoledronic acid
  Groups: Zoledronic acid
Drug: Any oral bisphosphonates marketed in Canada
  Groups: Oral Bisphosphonates

SUMMARY:
The study will assess the real life effectiveness of zoledronic acid in the management of patients with osteoporosis over 4 years of treatment. Zoledronic acid will be compared to oral bisphosphonates (OBP) with respect to the change in Bone Mineral Density (BMD) and incidence of fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patient is an ambulatory female 45 years of age or older
* Postmenopausal women with diagnosis of osteoporosis
* Prescription of zoledronic acid or any OBP as per the current Canadian monograph
* Must provide informed consent

Exclusion Criteria:

* Any prior use of iv bisphosphonates within the last 2 years
* Known secondary osteoporosis of any aetiology (hypogonadism in premenopausal women or premature menopause, malabsorption, chronic liver disease, inflammatory bowel disease)
* Metabolic bone diseases such as primary or secondary hyperparathyroidism, hypoparathyroidism, Paget's disease of bone, Fibrous dysplasia..
* Non-corrected hypocalcaemia at the time of zoledronic acid infusion
* Creatinine clearance < or = 30 ml/min
* Unwillingness or inability to comply with the study requirements
* Concurrent participation in a clinical trial of an investigational drug, or within the last 30 days

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ambulatory Female patients, at least 45 years of age, diagnosed with osteoporosis and taking either Zelodronic acid or any other oral bisphosphonates (OBP) as per the current Canadian monograph
Sampling Method: Non-Probability Sample
Enrollment: 1551 (Actual)
Dates: Start 2008-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Percent change in lumbar spine BMD as measured by dual energy x-ray absorptiometry (DXA) | 4 years

SECONDARY OUTCOMES:
change in femoral neck BMD as measured by dual energy x-ray absorptiometry (DXA) | 4 years
change in hip BMD as measured by dual energy x-ray absorptiometry (DXA) | 4 years
Percent change in hip BMD as measured by dual energy x-ray absorptiometry (DXA) | 4 years
Risk for fractures | 4 years
Burden of illness, health care resource utilization, and loss of productivity | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Marc Vaillancourt, Study Director — Novartis Pharmaceuticals Canada
Locations (3):
- Canada (3):
  - Vancouver, British Columbia
  - Hamilton, Ontario
  - Groupe de recherche en rhumatologie et maladies osseuses Inc, Québec, Quebec